CLINICAL TRIAL: NCT00001241
Title: Medical Therapy of Zollinger-Ellison Syndrome
Brief Title: Treatment of Zollinger-Ellison Syndrome
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 890015; 89-DK-0015
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-12-10

CONDITIONS: Zollinger Ellison Syndrome
Keywords: Gastric Acid Secretion; Histamine H2-Receptor Antagonists
MeSH Terms: conditions — Zollinger-Ellison Syndrome

SUMMARY:
In patients with Zollinger-Ellison Syndrome the level of gastric acid is elevated. This increased level of gastric acid is what causes the symptoms of the disease. Certain types of medication can control the secretion of gastric acid. In this study there are details on how drugs known as antihistamines (H2 receptor antagonists) can control the levels of gastric acid secretion.

The study describes; which patients are candidates for this research, what to do prior to initiating treatment, and the appropriate dose of antihistamine to be given.

Initial doses of the medication will be given intravenously (injected through a vein) and later doses will be administered orally (by mouth).

By following the procedure, researchers will be able to determine if there is a more effective route of drug administration, as well as the effectiveness of antihistamines in patients treated surgically for Zollinger-Ellison pancreatic tumors with mildly elevated gastric acid levels.

DETAILED DESCRIPTION:
This protocol describes the use of histamine H2-receptor antagonists to control gastric acid hypersecretion in patients with Zollinger-Ellison syndrome. It details which patients will be considered for treatment with these agents, the pretreatment procedures and the procedures to be followed in establishing the proper intravenous dose of histamine H2-receptor antagonist. It also details the procedure to be used to establish a safe and effective oral long-term maintenance dose of either cimetidine, ranitidine, nizatidine, or famotidine. By following these procedures it will be possible to evaluate the effectiveness of intravenous histamine H2 therapy if it is determined this is important for antisecretory control during periods when patients cannot take oral gastric antisecretory agents. It will also be possible to evaluate the effectiveness of histamine H2-receptor in patients with Zollinger-Ellison syndrome after successful gastrinoma resection who continue to have mild gastric hypersecretion.

ELIGIBILITY:
* INCLUSION CRITERIA:

Basal gastric acid secretion of greater than 15 mEq/hr (normal less than 10) or greater than 5 mEq/hr if they have had a previous gastric resection, a fasting plasma concentration of immunoreactive gastrin of greater than 100 pg/ml (normal less than 100), a positive secretin provocative tests or histological diagnosis of gastrinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1989-01-27; Study Completion 2007-12-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] McCarthy DM, Olinger EJ, May RJ, Long BW, Gardner JD. H2-Histamine receptor blocking agents in the Zollinger-Ellison syndrome. Experience in seven cases and implications for long-term therapy. Ann Intern Med. 1977 Dec;87(6):668-75. doi: 10.7326/0003-4819-87-6-668. PMID 22304